CLINICAL TRIAL: NCT05144711
Title: Selective Versus Nonselective Caries Excavation in Adults: Randomized Clinical Trial
Brief Title: Management of Deep Carious Lesions in Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 528/2021
Record Dates: First submitted 2021-11-22; First posted 2021-12-03 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Caries; Reversible Pulpitis
Keywords: Deep caries; Reversible pulpitis; Selective excavation; Nonselective excavation; Biodentine

STUDY DESIGN:
Intervention Model Description: Cases randomly assigned into the two groups using a block method
Who Masked: Participant, Outcomes Assessor
Masking Description: An informed consent will be obtained from the participant but he will not be informed whether selective or non selective excavation was done for him.
  the outcome assessor will be blinded to the procedure, and if required masking of the crowns of teeth on radiographs will be done before evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Selective excavation (Active Comparator): Cries will be removed from the peripheries of the cavity, while only soft caries will be removed from the plural side leaving stained leathery dentine that can not be removed by hand instruments. Biodentine will be placed and the cavity will be restored.
  Interventions: Procedure: Selective caries excavation
- Non selective excavation (Active Comparator): Caries will be cleaned form all cavity peripheries and floor. Biodentine will be placed and the toothy will be restored.
  Interventions: Procedure: Non selective caries excavation

INTERVENTIONS:
Procedure: Selective caries excavation — Selective caries excavation leaving stained but leathery dentine towards the pulp
  Arms: Selective excavation
Procedure: Non selective caries excavation — Complete excavation of caries regardless of the risk of pulp exposure
  Arms: Non selective excavation

SUMMARY:
Dental caries is one of the most prevalent non-communicable disease. However, despite its prevalence there is no consensus on how much caries to remove prior to placing a restoration to achieve optimal outcomes. Evidence for selective compared to complete nonselective excavation suggests there may be benefit for selective removal in sustaining tooth vitality while histological studies reveal that the remaining dentine is actually infected and may cause loss of vitality in long term.

The aim of this study is to randomly compare selective to non-elective excavation methods in carious mature permanent teeth with symptoms of reversible pulpitis

DETAILED DESCRIPTION:
The aim of this study is to randomly compare selective to nonselective excavation methods in carious mature permanent teeth with symptoms of reversible pulpitis over 4 years.

Cases will be collected from the initial treatment unit and the undergraduate clinics over a 8 months' period, the minimum sample size required is 120 teeth in 120 patients for an assumed difference of 20% in the success rate and accounting for 20% wear rate in the follow up, randomization will be performed using tabular randomization. Intensity of pulp symptoms will be recorded, patient's description of sensitivity to hot/cold/sweet lasting up to 15-20s and settling spontaneously are considered mild, while increased pain for more than several minutes and needing pain killers are considered severe.

Inclusion criteria:

* The patient age (16-60) years old
* Non -contributory medical history
* Deep caries extending>= 2/3 of dentine but not exposing the pulp on the radiograph
* The tooth should give positive response to cold testing
* Clinical diagnosis of reversible pulpitis
* The tooth is restorable, probing pocket depth and mobility are within normal limits
* No signs of pulpal necrosis including sinus tract or swelling
* No radiographic evidence of periapical changes indicative of apical periodontitis

Preoperative pulpal and periapical diagnosis will be established after clinical examination including soft tissue palpation, percussion, and cold testing (, and digital periapical and bitewing radiographs will be taken using film holders and a paralleling technique.

Baseline characteristics of the patient (age, gender) and the treated tooth (number, position, caries extension) will be recorded. Each tooth will be randomly allocated for the choice of treatment with selective or nonselective caries excavation according to a random sequence number generator.

Clinical procedure: The clinical procedure will be performed by one calibrated postgraduate student under supervision. The tooth will be anesthetized with , rubber dam will be applied and the tooth crown will be disinfected with 5% NaOCl before caries excavation; The cases will be divided randomly into:

Group 1: One-stage selective carious-tissue removal to soft or firm dentine, using carbon-steel rose- head burs (ash instruments) in a slow speed headpiece, the excavation end point is the detection of leathery dentine using a sharp dental explorer and excavator.

Group 2: Non-selective carious-tissue removal. The tooth will be isolated with rubber dam and disinfected with NaOCl. Complete caries excavation will be removed from the entire cavity, inspection under the microscope will be done to identify pulp exposure. If no pulp exposure is evident Biodentine will be placed and the cavity will be restored with composite. If pulp exposure occurred, and it is bleeding normally and uniformly red with no zones of degeneration or necrosis then direct pulp capping will be the choice of the treatment. The bleeding will be controlled via gentle pressure with a cotton pellet soaked with 2.5% NaOCl over the pulpal wound for 2 minutes and repeated if required up to 5 times.

In both groups, 2mm of Biodentine will be used and vitrebond will be placed as a liner on top, this will be followed by etching with 37% orthophosphoric acid, rinsing with water, and then bonding with adhesive followed by the placement of resin composite. Flowable composites will be used in deep cavities if needed. Clinical and radiographic success will be evaluated at 6 months, 1 year, 2 years and 4 years postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* The patient age (16-60) years old
* Non -contributory medical history
* Deep caries extending>= 2/3 of dentine but not exposing the pulp on the radiograph
* The tooth should give positive response to cold testing
* Clinical diagnosis of reversible pulpitis
* The tooth is restorable, probing pocket depth and mobility are within normal limits
* No signs of pulpal necrosis including sinus tract or swelling
* No radiographic evidence of periapical changes indicative of apical periodontitis

Exclusion Criteria:

* Immature roots
* caries exposing the pulp on radiograph
* symptoms of irreversible pulpits
* In ability to control bleeding after pulp exposure

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-10-03 (Actual); Primary Completion 2022-10-20 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Absence of clinical symptoms | 48 hours
  Relief of pain after the procedure

SECONDARY OUTCOMES:
Pulp vitality | 6, 12, 24, 48 months
  Absence of clinical and radiographic signs of pulp pathosis, in addition to normal response to cold testing

CONTACTS AND LOCATIONS:
Overall Officials: Nessrin Taha, PhD, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Jordan University of science and technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No
When recruitment is completed and the data is analyzed and submitted for publication. Data may be provided for the benefit of other researchers.

REFERENCES:
- [Result] Taha NA, About I, Sedgley CM, Messer HH. Conservative Management of Mature Permanent Teeth with Carious Pulp Exposure. J Endod. 2020 Sep;46(9S):S33-S41. doi: 10.1016/j.joen.2020.06.025. PMID 32950193
- [Derived] Taha NA, Ali MM, Abidin IZ, Khader YS. Pulp survival and postoperative treatment needs following selective vs. total caries removal in mature permanent teeth with reversible pulpitis: A randomized clinical trial. J Dent. 2024 Dec;151:105408. doi: 10.1016/j.jdent.2024.105408. Epub 2024 Oct 22. PMID 39442480